CLINICAL TRIAL: NCT04980209
Title: The Feasibility and Application of Intraoperative Ultrasound to Evaluate Femoral Head Shaping
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Cui Ligang, Chief Physician, Peking University Third Hospital
Other Study IDs: M2019453
Record Dates: First submitted 2021-07-02; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-06

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasonic and c-arm combination group: Ultrasound and c-arm were combined to evaluate intraoperatively conditions
  Interventions: Device: ultrasound evaluation
- c-arm group: c-arm group was used to evaluate intraoperatively conditions

INTERVENTIONS:
Device: ultrasound evaluation — According to the sequential test, the enrolled patients were divided into ultrasound evaluation group and no ultrasound evaluation group.
  Groups: Ultrasonic and c-arm combination group

SUMMARY:
To assess the feasibility of using intraoperative ultrasound to evaluate the femoral head formation; to evaluate the improvement of the forming effect using the intraoperative ultrasound combined with c-arm.

DETAILED DESCRIPTION:
Ultrasound can provide a multi-directional scan of the femoral head and neck junction, and the range of evaluation is larger than that of the intraoperative c-arm. The study was to assess the feasibility of using intraoperative ultrasound to evaluate the femoral head formation; to evaluate the forming of the femoral head and the improvement of the forming effect using the intraoperative ultrasound combined with c-arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip pain;
* Cam type (alpha Angle > 50°) impingement and glenoid labrum laceration

Exclusion Criteria:

* Previous hip surgery;
* Patients with subosseous cystic degeneration of synovitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the sequential test, the enrolled patients were divided into ultrasound evaluation group and no ultrasound evaluation group. Inclusion Criteria included patients with hip pain; Cam type (alpha Angle > 50°) impingement and glenoid labrum laceration.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
VAS scale | 1 year after operation
  Visual analogue scale（VAS）was used to measure the pain score. The minimum and maximum values were 0 and 10. The higher score, the worse pain.
MHHS scale | 1 year after operation
  Modified Harris Hip Score (MHHS) scale was used to measure the symptoms of joint. The minimum and maximum values were 0 and 91. The higher score, the better.
Hip CT | 1 day after operation
  Routine postoperative hip CT was used to understand the joint morphology.
Hip X-ray | 1 day after operation
  Routine hip X-ray at the Dunn position was conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Cui Ligang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking Univesity Third Hospital, Beijing, Beijing Municipality, China